CLINICAL TRIAL: NCT05874882
Title: Evaluating the Efficacy of Resveratrol Containing Mouthwash as Adjunct Treatment for Periodontitis:
Brief Title: Evaluating the Efficacy of Resveratrol Containing Mouthwash as Adjunct Treatment Periodontitis:
Acronym: resveratrol
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hadeel Mazin Akram, assistant professor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 744622
Record Dates: First submitted 2023-04-27; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Periodontitis
Keywords: mouthwash; periodontitis; resveratrol
MeSH Terms: conditions — Periodontitis | interventions — Root Planing; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: the study include three groups. one of them is the study group in which the patient will use resveratrol mouthwash as adjunct to scaling, the second group use chlorhexidine mouthwas as adjunct to scaling while the third group will use a placebo. all the participants and the examiner are blinded regarding the type of the mouthwash they will be using
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the supervisor will place the mouthwash in dark bottle with number so neither the examiner nor the patient will know the type of the mouthwash
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Placebo Comparator): patients with periodontitis will receive scaling and rootplaning and a placebo mouthwash twice daily for 4 weeks. saliva will be collected at the 1st visit and after one month then biochemical analysis for inflammatory biomarker will be done. periodontal parameters also will be evaluated at the 1st visit and after 1 month
  Interventions: Other: placebo mouthwash as adjunct to scaling and root planing in periodontitis patients
- chlorohexidine mouthwash (Active Comparator): patients with periodontitis will receive scaling and rootplaning and a chlorhexidine mouthwash twice daily for 4 weeks. saliva will be collected at the 1st visit and after one month then biochemical analysis for inflammatory biomarker will be done. periodontal parameters also will be evaluated at the 1st visit and after 1 month
  Interventions: Other: chlorhexidine mouthwash as adjunct to scaling and root planing in periodontitis patients
- resveratrol mouthwash (Experimental): patients with periodontitis will receive scaling and rootplaning and a resveratrol mouthwash twice daily for 4 weeks. saliva will be collected at the 1st visit and after one month then biochemical analysis for inflammatory biomarker will be done. periodontal parameters also will be evaluated at the 1st visit and after 1 month
  Interventions: Other: resveratrol mouthwash as adjunct to scaling and root planing in periodontitis patients

INTERVENTIONS:
Other: resveratrol mouthwash as adjunct to scaling and root planing in periodontitis patients — patients with periodontitis will receive scaling and rootplaning and a resveratrol mouthwash twice daily for 4 weeks. saliva will be collected at the 1st visit and after one month then biochemical analysis for inflammatory biomarker will be done. periodontal parameters also will be evaluated at the 1st visit and after 1 month
  Other Names: resveratrol mouthwash (oraxil)
  Arms: resveratrol mouthwash
Other: chlorhexidine mouthwash as adjunct to scaling and root planing in periodontitis patients — patients with periodontitis will receive scaling and rootplaning and a chlorhexidine mouthwash twice daily for 4 weeks. saliva will be collected at the 1st visit and after one month then biochemical analysis for inflammatory biomarker will be done. periodontal parameters also will be evaluated at the 1st visit and after 1 month
  Other Names: chlorhexidine mouthwash (corsodyl)
  Arms: chlorohexidine mouthwash
Other: placebo mouthwash as adjunct to scaling and root planing in periodontitis patients — patients with periodontitis will receive scaling and rootplaning and a placebo mouthwash twice daily for 4 weeks. saliva will be collected at the 1st visit and after one month then biochemical analysis for inflammatory biomarker will be done. periodontal parameters also will be evaluated at the 1st visit and after 1 month
  Other Names: placebo
  Arms: control

SUMMARY:
To evaluate the effectiveness of resveratrol mouthwash as adjunct to NSP treatment of periodontitis

DETAILED DESCRIPTION:
* Measuring and comparing the efficacy of RV mouth wash in comparison with CHX and placebo mouth wash in improving the clinical periodontal parameters;
* Measuring the salivary cytokines (IL-6) before and after 4weeks of the use of RV mouth wash as adjunct to NSP treatment in comparison with other mouthwash by using enzyme-linked immunosorbent assay.
* Measuring the salivary RANKL before and after 4weeks of the use of RV mouth wash as adjunct to NSP treatment in comparison with other mouthwash by using enzyme-linked immunosorbent assay.
* Correlate the salivary cytokines IL-6 and salivary RANKL with clinical periodontal parameter and with each other.
* Evaluate the intervention by using Visual analog scale (VAS)- score-based questionnaire will be filled out by each participant at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

-

The inclusion criteria:

1. Participants need to be systemically healthy with age > 18 years old.
2. Not taking antibiotic and anti-inflammatory drugs in the last three months.
3. At least 20 teeth should be present
4. Should have unstable periodontitis (PPD ≥ 5 or BOP at 4mm pocket)

The exclusion criteria:

1. Patients wearing fixed prosthesis (crowns, bridges or orthodontic appliances)
2. Those with chronic disease, immunocompromised patients, pregnant, on contraceptives or lactating women.
3. Those currently using any mouthwash.
4. Those on antibiotic therapy and anti-inflammatory medications during the study and in the last 3 months before the study.
5. Those having a history of hypersensitivity to any product used in the present study.
6. Those who are smokers or alcoholics.
7. Those who refuse to participate in the trial.

   -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
bleeding on probing | at1 month from the baseline
  bleeding on probing

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, Baghdad, None Selected, Iraq

IPD SHARING:
Plan to Share IPD: No